CLINICAL TRIAL: NCT03173937
Title: Unrelated Umbilical Cord Blood Transplantation for Severe Aplastic Anemia and Hypo-plastic MDS Using CordIn, Umbilical Cord Blood-Derived Ex Vivo Expanded Stem and Progenitor Cells, to Expedite Engraftment and Improve Transplant Outcome
Brief Title: Unrelated Umbilical Cord Blood Transplantation for Severe Aplastic Anemia and Hypo-plastic MDS Using CordIn(TM), Umbilical Cord Blood-Derived Ex Vivo Expanded Stem and Progenitor Cells to Expedite Engraftment and Improve Transplant Outcome
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 170091; 17-H-0091
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-28

CONDITIONS: Severe Aplastic Anemia; Hypo-Plastic MDS; Myelodysplastic Syndrome (MDS)
Keywords: Haploidentical; Nonmyeloablative
MeSH Terms: conditions — Anemia, Aplastic; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): CordIn is a cryopreserved stem/progenitor cell-based product of purified CD133+ cells composed of ex vivo expanded allogeneic UCB cells.
  Interventions: Biological: Omidubicel (former CordIn); Device: Miltenyi CliniMACS(R) CD34 Reagent System

INTERVENTIONS:
Biological: Omidubicel (former CordIn) — Stem/progenitor cell-based product of purified CD133+ cells composed of ex vivo expanded allogeneic umbilical/unrelated cord blood (UCB) cells. CordIn(TM) comprises: 1) cord blood-derived ex vivo expanded CD133+ cells (CordIn (TM) cultured fraction (CF)); and 2) the non-cultured cell fraction (CD133-) of the same CBU (CordIn(TM) Non-cultured Fraction (NF)). Both fractions, i.e. CordIn(TM) CF and CordIn(TM) NF are kept frozen until they are infused on the day of transplantation.
Device: Miltenyi CliniMACS(R) CD34 Reagent System — The CliniMACS CD34 Reagent System is a medical device system that is designed for the in vitro enrichment of CD34+ target cells from heterogeneous hematologic cell populations. The process of CD34+ cell selection results in simultaneous passive depletion of donor lymphocytes, potentially obviating the need for immunosuppressive drugs to prevent GVHD.

SUMMARY:
Background:

Severe aplastic anemia (SAA) and myelodysplastic syndrome (MDS) are bone marrow diseases. People with these diseases usually need a bone marrow transplant. Researchers are testing ways to make stem cell transplant safer and more effective.

Objective:

To test if treating people with SAA or MDS with a co-infusion of blood stem cells from a family member and cord blood stem cells from an unrelated donor is safe and effective.

Eligibility:

Recipients ages 4-60 with SAA or MDS

Donors ages 4-75

Design:

Recipients will be screened with:

* Blood, lung, and heart tests
* Bone marrow biopsy
* CT scan

Recipients will have an IV line placed into a vein in the neck. Starting 11 days before the transplant they will have several chemotherapy infusions and 1 30-minute radiation dose.

Recipients will get the donor cells through the IV line. They will stay in the hospital 3-4 weeks. After discharge, they will have visits:

* First 3-4 months: 1-2 times weekly
* Then every 6 months for 5 years

Donors will be screened with:

* Physical exam
* Medical history
* Blood tests

Donors veins will be checked for suitability for stem cell collection. They may need an IV line to be placed in a thigh vein.

Donors will get Filgrastim or biosimilar (G-CSF) injections daily for 5-7 days. On the last day, they will have apheresis: Blood drawn from one arm or leg runs through a machine and into the other arm or leg. This may be repeated 2 days or 2-4 weeks later.

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA) and myelodysplastic syndrome (MDS) are life-threatening bone marrow disorders. For SAA patients, long term survival can be achieved with immunosuppressive treatment. However, of those patients treated with immunosuppressive therapy, one quarter to one third will not respond, and about 50 percent of responders will relapse.

Combined haplo-cord transplant as an alternative to cord or haploidentical donor alone transplantation has recently been shown to be a viable transplant option for SAA patients lacking an HLA matched donor. In our ongoing protocol 08-H-0046, we have utilized this approach in 25 patients with SAA with 23/25 patients having sustained engraftment and long-term disease free/transfusion free survival. However, engraftment patterns have varied substantially and in some patients, cord engraftment was profoundly delayed or never occurred. A number of strategies to expand hematopoietic progenitor cells (HPC) in vitro to improve engraftment and prevent graft rejection have recently been studied. Nicotimanide (NAM) expanded umbilical cord blood/unrelated cord blood (UCB) can be successfully engrafted in NOD/SCID mice (1) and humans (2) where they appear to have long-term repopulating potential. CordIn(TM) is a cryopreserved stem/progenitor cell-based product of purified CD133+ cells composed of ex vivo expanded allogeneic UCB cells. CordIn(TM) comprises: 1) Ex vivo expanded, umbilical cord blood-derived hematopoietic CD34+ progenitor cells ( (CordIn(TM) cultured fraction (CF)); and 2) the non-cultured cell fraction of the same CBU (CordIn(TM) Non-cultured Fraction (NF)) consisting of mature myeloid and lymphoid cells. Both fractions, i.e. CordIn(TM) CF and CordIn(TM) NF are kept frozen until they are infused on the day of transplantation.

This research protocol is therefore designed to evaluate the safety and effectiveness of transplantation with ex vivo expanded UCB (CordIn(TM)) to overcome the high incidence of graft rejection associated with conventional UCB for aplastic anemia, where graft rejection occurs in up to 50% of subjects. We believe, based on preliminary data, that transplantation of CordIn(TM) will not only lead to rapid engraftment, but will also lead to sustained hematopoiesis, expedited immune recovery, and will reduce the chance of cord graft failure in this setting, potentially obviating the need for co-transplanting haploidentical CD34+ cells as a stem cell back-up. This phase II study is designed to have two cohorts: cohort 1 is intended to establish (in as safe a manner as possible) preliminary pilot data to support the capacity for the CordIn unit to engraft in patients with SAA in the presence of haplo CD34+ cells. For cohort 1, three to six subjects will be conditioned then will be transplanted with the thawed CordIn(TM) unit (consisting of the cultured fraction and the non-cultured fraction of the same CBU) and approximately 3 x 10^6 CD34+ cells/kg from a haploidentical donor which will serve as a backup stem cell source should cord graft failure occur. If 3 of the first 3 to 4 subjects or 4 of 6 subjects achieve early and sustained engraftment (defined as ANC >500 cells/ul by day 26 and a calculated cord ANC >500 cells /ul by day 42 sustained at day 100), the study will move to cohort 2 where up to 23 subsequent subjects will be transplanted with the CordIn(TM) unit alone.

The primary objective of the Phase II study is to evaluate the ability of the CordIn(TM) unit to achieve sustained early engraftment. Secondary endpoints will include 100 day and 200 day treatment related mortality (TRM), and standard transplant outcome variables such as non-hematologic toxicity, incidence and severity of acute and chronic GVHD, and relapse of disease. Health related quality of life will also be assessed as secondary outcome measure.

ELIGIBILITY:
* INCLUSION CRITERIA - RECIPIENT:
* Diagnosed with severe aplastic anemia with bone marrow cellularity <30% (excluding lymphocytes) associated with RBC or platelet transfusion dependence and/or neutropenia (absolute neutrophil count <=1000 cells/ uL or for patients receiving granulocyte transfusions, absolute neutrophil count <=1000 cells/ uL before beginning granulocyte transfusions).

OR

History of severe aplastic anemia transformed to MDS that meet the following criteria: a) International Prognostic Scoring System (IPSS) risk category of INT-1 or greater, b) < 5% myeloblasts and < 30% of cellularity in the bone marrow on screening morphologic analysis.

-Intolerance of or failure to respond to standard immunosuppressive therapy.

Identification of either a) at least one alternative donor (i.e. HLA- haploidentical related donor (i.e. >=5/10 HLA match: HLA-A, B, C, DR, and DQ loci) or >=9/10 HLA matched unrelated donor) who is available to serve as a stem cell donor for a salvage allogeneic transplant in the event that the CordIn(TM) unit has been rejected or b) umbilical cord blood unit/s that can be used for a salvage cord blood transplant in the event that the CordIn(TM) unit has been rejected.

-Availability of at least one >=4/8 HLA matched (HLA-A, B, C, and DR loci) cord blood unit from the National Marrow Donor Program (NMDP).

The cord blood unit must contain a minimum TNC of at least 1.8 x 10^9 and at least 1.5x10^7/kg TNC and at least 8 x 10^6 CD34+ cells (all doses prior to thawing).

Exception: Cord units containing at least 8 x 10^6 CD34+ cells but less than 1.8 x 10^9 TNC may be eligible for use on this trial if

1. the pre-expansion CD34/kg recipient cell number is at least 1.5 x 10^5 /kg

   AND
2. approval for use of this cord unit for expansion is granted by Gamida Cell.
3. the final cell counts on the cultured and non-cultured fractions meet the IND specified minimal release criteria.

   * The CBU will have undergone volume reduction (both plasma and red blood cell depletion) prior to cryopreservation. All CBUs should be procured from public banks that meet local applicable regulations.
   * Ages 4-60 years inclusive.
   * Ability to comprehend the investigational nature of the study and provide informed consent. The procedure will be explained to subjects aged 4-17 years with formal consent being obtained from parents or legal guardian.

EXCLUSION CRITERIA - RECIPIENT (ANY OF THE FOLLOWING):

* Availability of an HLA identical (12/12) matched related or unrelated donor who is available within optimal timeline and suitable considering graft source and established donor selection factors (e.g. age, sex, viral exposure, ABO compatibility, pregnancy status, etc) per PI discretion.
* ECOG performance status of 2 or more.
* Major anticipated illness or organ failure incompatible with survival from transplant.
* Current pregnancy, or unwillingness to take oral contraceptives or use a barrier method of birth control or practice abstinence to refrain from pregnancy, if of childbearing potential for one year.
* HIV positive.
* Diagnosis of Fanconi s anemia (by chromosome breakage study).
* Diffusion capacity of carbon monoxide (DLCO) <40% using DLCO corrected for Hgb or lung volumes (patients under the age of 10 may be excluded from this criterion if they have difficulty performing the test correctly and thus are unable to have their DLCO assessed).
* Left ventricular ejection fraction < 40% (evaluated by ECHO).
* Transaminases > 5x upper limit of normal.
* Serum bilirubin >4 mg/dl.
* Creatinine clearance < 50 cc/min/BSAm2 by 24-hour urine collection adjusted by body surface area.
* Serum creatinine > 2.5 mg/dl
* Presence of an active infection not adequately responding to appropriate therapy.
* History of a malignant disease liable to relapse or progress within 5 years.
* Allergy to bovine, Gentamicin, or to any product which may interfere with the treatment.
* Presence of donor-specific antibodies (DSA) to the umbilical cord blood unit and for cohort 1, to the haplo-identical donor.

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2017-06-13 (Actual); Primary Completion 2027-04-28 (Estimated); Study Completion 2032-03-01 (Estimated)

PRIMARY OUTCOMES:
Cord engraftment | At or before day 100
  Cord engraftment

SECONDARY OUTCOMES:
Treatment related mortality (TRM), and standard transplant outcome variables such as non-hematologic toxicity, incidence and severity of acute and chronic GVHD, and relapse of disease | 100 day and 200 day
  treatment related mortality

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Childs, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-H-0091.html